CLINICAL TRIAL: NCT02764190
Title: Delivering Patient-Centered Adolescent Preventative Care With Training and Technology
Brief Title: I-ACT With Check Yourself
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Carolyn McCarty, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IHS-1402-10592
Record Dates: First submitted 2016-04-29; First posted 2016-05-06 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- I-ACT with Check Yourself (Experimental): Adolescents complete Check Yourself which delivers personalized, motivational feedback on their health behaviors prior to their primary care appointment. Check Yourself includes the provision of age normative feedback, goal setting strategies, and strategies to highlight discrepancies. Primary care providers will receive I-ACT and the Check Yourself summary report of health risk behaviors before an adolescent patient's appointment. I-ACT will provide training in adolescent-preferred communication methods and use of Check Yourself as a framework for the provider to use motivational interviewing to consider the patients' change readiness and their personal health goals. I-ACT includes online interactive, case-based learning, with booster sessions and feedback reports to reinforce new skills.
  Interventions: Behavioral: I-ACT with Check Yourself
- Usual care (No Intervention): In the usual care group, adolescents are asked to complete health risk screening on a computer. No personalized feedback is provided to adolescents and primary care providers do not receive I-ACT or the Check Yourself summary report of the adolescent's health risk behaviors.

INTERVENTIONS:
Behavioral: I-ACT with Check Yourself
  Arms: I-ACT with Check Yourself

SUMMARY:
Adolescents have some of the highest rates of risk behaviors of all age groups and health behaviors developed in adolescence can persist into adulthood. These behaviors carry significant risks for subsequent disease, disability, and healthcare burden. Despite these risks, health risk screening in primary care is infrequently performed and results are rarely followed by targeted intervention. In response to the need for screening-linked interventions, our study team has developed a web-based, electronic Personalized Motivational Feedback tool which we refer to as "Check Yourself." Based on motivational interviewing, a technique to mobilize personal change, Check Yourself is designed to promote healthy choices for the multiple behaviors relevant to adolescents as well as to provide information to providers to promote discussions around health behaviors between providers and adolescents.

Building on electronic health interventions, primary care providers can play an essential role in helping adolescents to make healthy behavior choices. Emerging evidence suggests that the consistency of preventive counseling can be increased through provider training and the provision of screening tools; yet, we know very little about the quality of such counseling, and if it impacts outcomes that are important to adolescent patients themselves.

This study is a stepped-wedge, controlled trial comparing the effectiveness of an interactive adolescent-centered training for primary care providers (I-ACT) and Check Yourself to usual care. This study will take place in six pediatric practices. The purpose of this study is to determine whether this system of interventions (i.e., I-ACT, Check Yourself, and the summary report) is more effective than usual care in reducing health risk behaviors, improving adolescent motivation for health, and improving quality of care among adolescents receiving primary health care services.

ELIGIBILITY:
Inclusion Criteria:

* Eligible adolescent participants will be 13-18 years of age and caregiver participants will be 18 years of age or older and able to understand English. Eligible participants will have an appointment (or have a child with an appointment) with a participating medical practice.

Exclusion Criteria:

* Adolescents will be excluded from the study if they do not meet age requirements, do not have an appointment with a participating provider at a PSPRN clinic, lack the means to complete follow-up interviews (i.e., have neither telephone nor internet access), have a sibling who has been/is being enrolled in the study or have previously participated in our previous trial comparing Check Yourself to usual care, and/or are not able to understand English.
* Caregivers will be excluded from the study if they do not speak English; or if their child is not eligible or declines to participate in the study .

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 302 (Actual)
Dates: Start 2016-10; Primary Completion 2018-02 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] McCarty CA, Parker E, Zhou C, Katzman K, Stout J, Richardson LP. Electronic Screening, Feedback, and Clinician Training in Adolescent Primary Care: A Stepped-Wedge Cluster Randomized Trial. J Adolesc Health. 2022 Feb;70(2):234-240. doi: 10.1016/j.jadohealth.2021.07.019. Epub 2021 Aug 14. PMID 34404610

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: I-ACT With Check Yourself: Adolescents completed Check Yourself which delivered personalized, motivational feedback to them on their health behaviors prior to their primary care appointment. Primary care providers received training (I-ACT) and the Check Yourself summary report of health risk behaviors before the adolescent's appointment. I-ACT consisted of online, interactive training in adolescent-preferred communication methods and motivational interviewing, with booster sessions and feedback reports to reinforce new skills.
- No Intervention: Usual Care: In the usual care group, adolescents are asked to complete health risk screening on a computer. No personalized feedback is provided to adolescents and primary care providers do not receive I-ACT or the Check Yourself summary report of the adolescent's health risk behaviors.
Period: Overall Study
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Started | 167 | 135
1 Day Follow-up | 161 | 131
3 Month Follow-up | 156 | 128
6 Month Follow-up | 155 | 128
12 Month Follow-up | 150 | 122
Completed | 150 | 122
Not Completed | 17 | 13
Not completed — Lost to Follow-up | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care | Total
Number analyzed (Participants) | 167 | 135 | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 167 | 135 | 302
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.79 (1.41) | 14.70 (1.44) | 14.75 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 69 | 157
  Male | 79 | 66 | 145
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 2 | 4 | 6
  Native American | 0 | 1 | 1
  Asian | 11 | 17 | 28
  Caucasian | 122 | 90 | 212
  Hispanic | 11 | 6 | 17
  Other/Multiple Races | 21 | 17 | 38
Region of Enrollment [Number; unit: participants]
  United States | 167 | 135 | 302

OUTCOME MEASURES:

1. Primary Outcome: Number of Health Risk Behaviors
Description: The risk behavior scale includes 22 values: 0 (min) to 21 (max). Higher scores indicate a worse outcome. Endorsement of any of the following counts as 1 (moderate risk) or 2 (high risk) on the scale depending on response and participant: ≥2 sugar-sweetened beverages consumed during typical day; ≤3 servings fruits/vegetables consumed during typical day; ≤3 days with 60+ minutes exercise during typical week; texting while driving in past 3 months; ≤7 hrs of sleep during typical night; not "always" using seatbelt; not "always" using helmet when bicycling; having driven under the influence of substances; tobacco use; days alcohol consumption in last 30 days (risk based on age) and/or number of drinks per drinking episode (risk based on age & sex); days marijuana consumption in last 30 days (risk based on age) and/or other drug use in past 3 months; not using birth control during last sexual intercourse and/or not "always" using a condom; & score of ≥10 on PHQ-9 depression.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 150 | 120
score on a scale | 2.23 (1.98) | 2.62 (2.02)

2. Primary Outcome: Sweetened Beverage Consumption
Description: Adolescent self-reported number of sweetened beverages consumed in a typical day in the past 3 months. The sweetened beverages scale includes 4 values: 0 (min), 1, 2, or 3+ (max) sweetened beverages per day. Higher scores mean a worse outcome.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 0.80 (0.80) | 0.95 (1.05)

3. Primary Outcome: Fruit and Vegetable Consumption
Description: Adolescent self-reported number of fruits and vegetables consumed in a typical day in the past 3 months. The fruits and vegetables scale includes 6 values: 0 (min), 1, 2, 3, 4, or 5+ (max). Higher scores mean a better outcome.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 127
score on a scale | 2.84 (1.29) | 2.53 (1.17)

4. Primary Outcome: Physical Activity
Description: Adolescent self-reported number of days with >60 minutes of physical activity in an average week in the past 3 months. The physical activity scale includes 8 values: 0 (min) to 7 (max). Higher scores mean a better outcome.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 126
score on a scale | 4.81 (1.72) | 4.26 (1.66)

5. Primary Outcome: Sleep
Description: Adolescent self-reported hours of sleep on a typical night in the past 3 months. The sleep scale includes 13 values: 0 (min) to 12+ (max) hours of sleep per night. Higher scores mean a better outcome.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 152 | 124
score on a scale | 7.75 (1.26) | 7.73 (1.39)

6. Primary Outcome: Alcohol Consumption (Frequency)
Description: Adolescent self-reported number of days of alcohol consumption in the past month. Alcohol frequency scale includes 31 values: 0 (min) to 30 (max) days in the past month. Higher scores mean a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 0.25 (1.09) | 0.25 (1.28)

7. Primary Outcome: Alcohol Consumption (Quantity)
Description: Adolescent self-reported number of drinks during a typical drinking episode in the prior month. The alcohol quantity scale includes 16 values from 0 (min) to 15+ (max). Higher score means a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 0.20 (0.79) | 0.10 (0.53)

8. Primary Outcome: Marijuana Consumption
Description: Adolescent self-reported number of days using marijuana in the past month. The marijuana frequency scale includes 31 values: 0 (min) to 30 (max) days in the past month. Higher scores mean a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 0.53 (3.05) | 0.14 (0.97)

9. Primary Outcome: Other Drug Consumption
Description: Adolescent self-reported use of other drugs in the past 3 months. The other drug score includes 2 values: 0=no (min) and 1=yes (max). Higher scores mean a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 0.02 (0.14) | 0.00 (0.00)

10. Primary Outcome: Depression
Description: Adolescent self-reported depression as measured on the nine item Patient Health Questionnaire (PHQ-9) in the past 2 weeks. The PHQ-9 depression scale includes 28 values: 0 (min) to 27 (max). Higher scores mean a worse outcome.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 3.02 (4.14) | 3.41 (4.16)

11. Primary Outcome: Seatbelt Use
Description: Adolescent self-reported frequency of seatbelt use in a car in the past 3 months. The seatbelt use scale includes 4 values: 1=never (min), 2=sometimes, 3=usually, or 4=always (max). Higher scores mean a better outcome.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 3.97 (0.18) | 3.94 (0.24)

12. Primary Outcome: Helmet Use
Description: Adolescent self-reported frequency of helmet use while bicycling in the past 3 months. The helmet use scale includes 4 values: 1=never (min), 2=sometimes, 3=usually, or 4=always (max). Higher scores mean a better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 153 | 128
score on a scale | 3.78 (0.69) | 3.52 (1.0)

13. Primary Outcome: Texting While Driving
Description: Adolescent self-reported endorsement of texting while driving in the past 3 months. This question is only asked among adolescents who drive a car. The texting while driving scale includes 4 values: 1=never (min), 2=sometimes, 3=usually, or 4=always (max). Higher scores mean a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 1.06 (0.24) | 1.07 (0.26)

14. Primary Outcome: Condom and/or Birth Control Use
Description: Adolescent self-reported condom use with sexual intercourse in the past 3 months and/or use of birth control at last sexual intercourse. Two questions were used for this category. These questions were asked only to sexually active youth. The condom use scale includes 4 values: 1=always (min), 2=often, 3=sometimes, 4=never (max). Higher scores mean a worse outcome. The birth control scale includes 2 values: 0=no (min), 1=yes (max). Higher scores mean a better outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 9 | 3
score on a scale
  Condom Use | 1.89 (1.36) | 2.00 (1.0)
  Birth Control Use | 1.0 (0.00) | 1.0 (0.0)

15. Primary Outcome: Driving With Impairment
Description: Adolescent self-reported driving under the influence of a substance in the past 3 months. This question was asked only of adolescents who drive a car. The driving with impairment scale includes 2 values: 0=no (min) and 1=yes (max). Higher scores mean a worse outcome.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 0.01 (0.08) | 0.02 (0.13)

16. Primary Outcome: Adolescent Satisfaction With Care
Description: Adolescent satisfaction with care is assessed using one item adapted from the Consumer Assessment of Healthcare Providers and Systems (CAHPS) measure at 1-day follow-up. The CAHPS scale includes 10 values: 1 (min) to 10 (max). Higher scores mean a better outcome.
Time Frame: 1-day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 148 | 119
score on a scale | 9.18 (1.11) | 9.23 (0.95)

17. Primary Outcome: Caregiver Satisfaction With Care
Description: Caregiver satisfaction with care is assessed using the four items adapted from the Consumer Assessment of Healthcare Providers and Systems (CAHPS) measure at 1-day follow-up. Scores on this scale range from 3 (min) to 22 (max) with higher scores indicating higher satisfaction with care.
Time Frame: 1-day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 115 | 100
score on a scale | 21.54 (0.76) | 21.47 (1.13)

18. Primary Outcome: Adolescent Perception of Patient-Centeredness
Description: The total score on the Consultation and Relational Empathy measure (CARE) is used to assess adolescent self-report of perceived patient-centeredness from their primary care provider. Scores on the scale range from 10 (min) to 50 (max) with higher scores indicating a better outcome.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 150 | 123
score on a scale | 45.63 (5.60) | 45.63 (6.26)

19. Primary Outcome: Tobacco Use
Description: Adolescent self-reported tobacco use in the past 3 months. The tobacco use scale includes 2 values: 0=no (min) or 1=yes (max). Higher scores mean a worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 154 | 128
score on a scale | 0.03 (0.16) | 0.02 (0.13)

20. Secondary Outcome: Percent of Risk Behaviors Counseled on During Primary Care Appointment
Description: Percent of adolescent-reported health risk behaviors discussed with the healthcare provider during the primary care visit adjusted for the total number of health risk behaviors reported at baseline.
Time Frame: 1 day
Measure: Number; unit: percentage of risk behaviors counselled
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
Number analyzed (Participants) | 152 | 123
percentage of risk behaviors counselled
  Moderate risk behaviors | 43 | 35
  High risk behaviors | 36 | 23

21. Secondary Outcome: Number of Health Risk Behaviors
Description: Adolescent total count health-risk behaviors at 6 month follow-up including: During typical day: ≥2 sugar-sweetened beverages consumed and ≤3 servings fruits/vegetables consumed; ≤3 days with 60+ minutes exercise during typical week; having texted while driving in past 3 months; ≤7 hours of sleep during typical night; not "always" using seatbelt; not "always" using helmet when bicycling; having driven under the influence of substances; tobacco use; days of alcohol consumption in last 30 days (risk based on age: ≥1 day/30 days (ages 13-15), ≥2 days/30 days (ages 16-17), or ≥3 days/30 days (age 18))and/or number of drinks per drinking episode (risk based on age and sex: ≥3 (Girls 13-17; Boys 13), ≥4 (Girls 18; Boys 14-15), or ≥5 (Boys 16-18)); days marijuana consumption in 30 day (risk based on age) and/or other drugs use in past 3 months; not using birth control during last sexual intercourse and/or not "always" using a condom; and score of ≥10 on PHQ-9.
Time Frame: 6 month
Reporting Status: Not Posted

22. Secondary Outcome: Number of Health Risk Behaviors
Description: Adolescent total count health-risk behaviors at 12 month follow-up including: During typical day: ≥2 sugar-sweetened beverages consumed and ≤3 servings fruits/vegetables consumed; ≤3 days with 60+ minutes exercise during typical week; having texted while driving in past 3 months; ≤7 hours of sleep during typical night; not "always" using seatbelt; not "always" using helmet when bicycling; having driven under the influence of substances; tobacco use; days of alcohol consumption in last 30 days (risk based on age: ≥1 day/30 days (ages 13-15), ≥2 days/30 days (ages 16-17), or ≥3 days/30 days (age 18))and/or number of drinks per drinking episode (risk based on age and sex: ≥3 (Girls 13-17; Boys 13), ≥4 (Girls 18; Boys 14-15), or ≥5 (Boys 16-18)); days marijuana consumption in 30 day (risk based on age) and/or other drugs use in past 3 months; not using birth control during last sexual intercourse and/or not "always" using a condom; and score of ≥10 on PHQ-9.
Time Frame: 12 month
Reporting Status: Not Posted

23. Secondary Outcome: Sweetened Beverage Consumption
Description: Adolescent self-reported sweetened beverages consumed in a typical day in past 3 months
Time Frame: 6 month
Reporting Status: Not Posted

24. Secondary Outcome: Sweetened Beverage Consumption
Description: Adolescent self-reported sweetened beverages consumed in a typical day in past 3 months
Time Frame: 12 month
Reporting Status: Not Posted

25. Secondary Outcome: Fruit and Vegetable Consumption
Description: Adolescent self-reported fruits and vegetables consumed in a typical day in past 3 months
Time Frame: 6 month
Reporting Status: Not Posted

26. Secondary Outcome: Fruit and Vegetable Consumption
Description: Adolescent self-reported fruits and vegetables consumed in a typical day in past 3 months
Time Frame: 12 month
Reporting Status: Not Posted

27. Secondary Outcome: Physical Activity
Description: Adolescent self-reported days with >60 minutes of physical activity in an average week in past 3 months
Time Frame: 6 month
Reporting Status: Not Posted

28. Secondary Outcome: Physical Activity
Description: Adolescent self-reported days with >60 minutes of physical activity in an average week in past 3 months
Time Frame: 12 month
Reporting Status: Not Posted

29. Secondary Outcome: Sleep
Description: Adolescent self-reported hours of sleep on a typical night in past 3 months
Time Frame: 6 month
Reporting Status: Not Posted

30. Secondary Outcome: Sleep
Description: Adolescent self-reported hours of sleep on a typical night in past 3 months
Time Frame: 12 month
Reporting Status: Not Posted

31. Secondary Outcome: Alcohol Consumption
Description: Adolescent self-reported number of days of alcohol consumption and drinks during typical drinking episode in the prior month
Time Frame: 6 month
Reporting Status: Not Posted

32. Secondary Outcome: Alcohol Consumption
Description: as for outcome 31
Time Frame: 12 month
Reporting Status: Not Posted

33. Secondary Outcome: Marijuana and/or Other Drug Consumption
Description: Adolescent self-reported number of days using marijuana in the past month and/or other drugs used in past 3 months
Time Frame: 6 month
Reporting Status: Not Posted

34. Secondary Outcome: Marijuana and/or Other Consumption
Description: Adolescent self-reported number of days using marijuana in the past month and/or other drugs used in past 3 months
Time Frame: 12 month
Reporting Status: Not Posted

35. Secondary Outcome: Depression
Description: Adolescent self-reported depression as measured on the nine item Patient Health Questionnaire in past 2 weeks
Time Frame: 6 month
Reporting Status: Not Posted

36. Secondary Outcome: Depression
Description: Adolescent self-reported depression as measured on the nine item Patient Health Questionnaire in past 2 weeks
Time Frame: 12 month
Reporting Status: Not Posted

37. Secondary Outcome: Seatbelt Use
Description: Adolescent self-reported frequency of seatbelt use in a car in past 3 months
Time Frame: 6 month
Reporting Status: Not Posted

38. Secondary Outcome: Seatbelt Use
Description: Adolescent self-reported frequency of seatbelt use in a car in past 3 months
Time Frame: 12 month
Reporting Status: Not Posted

39. Secondary Outcome: Helmet Use
Description: Adolescent self-reported frequency of helmet use while bicycling in past 3 months
Time Frame: 6 month
Reporting Status: Not Posted

40. Secondary Outcome: Helmet Use
Description: Adolescent self-reported frequency of helmet use while bicycling in past 3 months
Time Frame: 12 month
Reporting Status: Not Posted

41. Secondary Outcome: Texting While Driving
Description: Adolescent self-reported endorsement of texting while driving in past 3 months
Time Frame: 6 month
Reporting Status: Not Posted

42. Secondary Outcome: Texting While Driving
Description: Adolescent self-reported endorsement of texting while driving in past 3 months
Time Frame: 12 month
Reporting Status: Not Posted

43. Secondary Outcome: Condom Use and/or Birth Control Use
Description: Adolescent self-reported condom use with sexual intercourse in the past 3 months and/or use of birth control at last sexual intercourse
Time Frame: 6 month
Reporting Status: Not Posted

44. Secondary Outcome: Condom Use and/or Birth Control Use
Description: as for outcome 43
Time Frame: 12 month
Reporting Status: Not Posted

45. Secondary Outcome: Driving With Alcohol Impairment
Description: Adolescent self-reported driving under the influence of a substance
Time Frame: 6 month
Reporting Status: Not Posted

46. Secondary Outcome: Driving With Alcohol Impairment
Description: Adolescent self-reported driving under the influence of a substance
Time Frame: 12 month
Reporting Status: Not Posted

47. Secondary Outcome: Interval Receipt of Care Questionnaire
Description: Dichotomous variable indicating receipt of any follow-up care to address risk behaviors identified at baseline adjusted for baseline number of health risk behaviors.
Time Frame: 3 month
Reporting Status: Not Posted

48. Secondary Outcome: Interval Receipt of Care Questionnaire
Description: Dichotomous variable indicating receipt of any follow-up care to address risk
Time Frame: 6 month
Reporting Status: Not Posted

49. Secondary Outcome: Interval Receipt of Care Questionnaire
Description: Dichotomous variable indicating receipt of any follow-up care to address risk
Time Frame: 12 month
Reporting Status: Not Posted

50. Secondary Outcome: Readiness to Change Ruler Questionnaire
Description: Assessment of adolescent reported motivation to change overall health using a Readiness to Change Ruler.
Time Frame: 1 day
Reporting Status: Not Posted

51. Secondary Outcome: Readiness to Change Ruler Questionnaire
Description: Assessment of adolescent reported motivation to change overall health using a Readiness to Change Ruler.
Time Frame: 3 month
Reporting Status: Not Posted

52. Secondary Outcome: Readiness to Change Ruler Questionnaire
Description: Assessment of adolescent reported motivation to change overall health using a Readiness to Change Ruler.
Time Frame: 6 month
Reporting Status: Not Posted

53. Secondary Outcome: Readiness to Change Ruler Questionnaire
Description: Assessment of adolescent reported motivation to change overall health using a Readiness to Change Ruler.
Time Frame: 12 month
Reporting Status: Not Posted

54. Secondary Outcome: Tobacco Use
Description: Adolescent self-reported tobacco use in past 3 months
Time Frame: 6 month
Reporting Status: Not Posted

55. Secondary Outcome: Tobacco Use
Description: Adolescent self-reported tobacco use in past 3 months
Time Frame: 12 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 3 months.
Arm/Group | Experimental: I-ACT With Check Yourself | No Intervention: Usual Care
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/135
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/135
Other Adverse Events (participants affected / at risk) | 0/167 | 0/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT02764190/Prot_SAP_000.pdf